CLINICAL TRIAL: NCT06189105
Title: Testing the Efficacy and Safety of Niacinamide Cosmetic Preparation: A Randomised, Controlled Trial
Brief Title: Efficacy and Safety Assessment of Niacinamide Cosmetic Preparation: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Dario Leskur, assistant professor, University of Split, School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2181-198-03-04-23-032
Record Dates: First submitted 2023-09-13; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Skin Hyperpigmentation; Dry Skin; Eczema
MeSH Terms: conditions — Hyperpigmentation; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): Use of facial serum with
  niacinamide, plant-based collagen and
  peptides on randomized site on forehead
  Interventions: Other: miss alice face it you love me serum
- placebo comparator (Placebo Comparator): No treatment (usual
  skincare rutine)
  Interventions: Other: No treatment (usual skincare rutine)

INTERVENTIONS:
Other: miss alice face it you love me serum — Facial serum with niacinamide, plant-based collagen and peptides will be applied by each participant to the treatment site according to randomization protocol every evening
  Arms: experimental arm
Other: No treatment (usual skincare rutine) — No treatment (usual skincare rutine)
  Arms: placebo comparator

SUMMARY:
Niacinamide in lower concentrations has been recognized as a cosmetic ingredient with hydrating properties. Therefore, aim was to test the efficacy and safety of niacinamide cosmetic preparation in A Randomized, Controlled Trial.

DETAILED DESCRIPTION:
Skin hydration (as use of hydrating cosmetic ingredients) is one of the most interventions for healthy skin and skin barrier function. Therefore, cosmetic ingredients used for this purpose should be examined for their efficacy.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers who gave written informed consent

Exclusion Criteria:

* skin disease, skin damage on measurement sites, use of corticosteroids and immunomodulators a month prior to the inclusion and during the trial, non-adherence to the trial protocol, exposure to artificial UV radiation, pregnancy and lactation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
TEWL assessment with Courage Khazaka probe | through study completion, an average of 1 year
  Transepidermal water loss
Hydration assessment with corneometer probe | through study completion, an average of 1 year
  stratum corneum hydration
pigmentation assessment with mexameter probe | through study completion, an average of 1 year
  erythema and melanin
skin oiliness assessment with sebumeter probe | through study completion, an average of 1 year
  sebum level

SECONDARY OUTCOMES:
subjective opinion of participants | through study completion, an average of 1 year
  participants notes on skin rection

CONTACTS AND LOCATIONS:
Overall Officials: Dario Leskur, Study Director — USSM
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Yes
upon request
Supporting Information: CSR
Time Frame: upon request
Access Criteria: upon request

REFERENCES:
- [Derived] Rusic D, Ivic M, Slugan A, Leskur D, Modun D, Durdov T, Vukovic D, Bukic J, Bozic J, Seselja Perisin A. Pilot Study on the Effects of a Cosmetic Serum Containing Niacinamide, Postbiotics and Peptides on Facial Skin in Healthy Participants: A Randomized Controlled Trial. Life (Basel). 2024 Dec 18;14(12):1677. doi: 10.3390/life14121677. PMID 39768384